CLINICAL TRIAL: NCT03437486
Title: Mechanisms of Familial Pulmonary Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Margaret Salisbury, Dr. Margaret Salisbury, Vanderbilt University Medical Center
Other Study IDs: 080780
Record Dates: First submitted 2017-06-16; First posted 2018-02-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Familial Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Familial Interstitial Pneumonia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, including DNA, plasma and serum, along with BAL fluid and transbronchial biopsies will be collected and used for biomarker studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Familial Pulmonary Fibrosis: Subjects asked to participate in this study will be unaffected family members of patients previously diagnosed with familial interstitial pneumonia (FIP) which is the familial form of idiopathic pulmonary fibrosis (IPF).

SUMMARY:
This a prospective, longitudinal study of first-degree family members of patients diagnosed with familial interstitial pneumonia (FIP). FIP is the familial form of idiopathic pulmonary fibrosis (IPF), which is defined as 2 or more bloodline relatives which have a diagnosis of idiopathic interstitial pneumonia (IIP). The most common form of idiopathic interstitial pneumonia in FIP families is IPF (approximately 70%). The inheritance pattern in FIP is consistent with autosomal dominant inheritance with incomplete penetrance. Therefore, individuals in this study have approximately 50% risk of carrying a disease-associated allele. The causative gene is currently only known approximately 20% of families. The main goal of this longitudinal study is to better establish the natural history of FIP and to identify risk factors for later development of symptomatic disease. The investigators' plan is to follow these at-risk individuals with yearly questionnaires and planned in person 2 year follow-ups through age 75 or until they develop symptomatic FIP.

DETAILED DESCRIPTION:
Potential research subjects will be sent a questionnaire (modified version of the ATS-DLD-78 questionnaire) and study consent form. Individuals with no prior history of lung disease and a dyspnea score of 2 or less will be offered the opportunity to undergo further research evaluation, which will include HRCT scanning, pulmonary function testing (PFTs) and blood draw. During the years 2024-2029, these visits will also contain an additional questionnaire, a urine specimen, and the use of wearable devices to further investigate the environmental factors that may contribute to pulmonary fibrosis. Subjects with grade 3 or greater dyspnea or findings of extensive disease on HRCT scan (see below), will be recommended to undergo clinical diagnostic evaluation outside the study. For those subjects that participate in this study, demographic information will be collected and stored in a database, including past medical history, smoking history, medications, and occupational and environmental exposure history.

Approximately every 3 years, we may contact you to return to Vanderbilt for another round of blood draw, high resolution CT scan of your lungs, and Pulmonary Function Tests (PFTs). These tests are repeated to help us understand whether changes in blood, CT scan, or lung function can predict the development of pulmonary fibrosis in relatives of patients with pulmonary fibrosis. We expect the follow-up period to last approximately 10 years (from the first study visit). Subjects will be asked to complete no more than 6 total blood/HRCT/PFT collections.

Each year after enrollment, the investigators will perform follow-up to ascertain whether subjects have: 1) developed respiratory symptoms consistent with FIP/IPF, 2) undergone additional diagnostic evaluations for lung disease, or 3) begun any new treatments for lung disease. Subjects who have developed respiratory symptoms will be encouraged to seek medical evaluation. For those who have undergone any new diagnostic testing or have been diagnosed with FIP, study coordinators will seek permission to obtain HRCTs, medical records, pulmonary function test results, and lung blocks for evaluation by investigators in this study.

The investigators will use standard criteria established by the ATS/ERS to guide the diagnostic classification of patients who develop FIP. Information will be reviewed by a pathologist, a radiologist, and 3 clinicians. In all cases, the clinicians make the final diagnosis and after reviewing the clinical material (clinical/demographic data and pulmonary physiology), and the radiology and pathology data.

HRCT: A single prone HRCT scan without intravenous contrast will be performed and read by an expert chest radiologist. He will assess the presence, extent, and distribution of areas of ground-glass attenuation, interlobular reticular opacities, irregular thickening of interlobular septa, traction bronchiectasis, and traction bronchiolectasis. The anatomic distribution of each finding will be classified in each lung in one of 4 zones from apex to base (upper, middle, lower, lowest). A score of 0 (absent), 1 (<5%), or 2 (>5% parenchymal involvement) will be given for each descriptor in each lung zone based on visual estimation (total score of 1-16). In addition, HRCT scans will be classified as: 1) normal, 2) abnormal, consistent with early FIP, 3) abnormal, consistent with extensive disease, or 4) abnormal, consistent with other diagnoses. Extensive disease is defined as >5% honeycombing in >2 zones. Other diagnoses could include suspicious lung nodules, extensive emphysema, or other findings requiring clinical referral. Disease progression on HRCT is defined by an increase in the total CT score.

Pulmonary function testing: PFTs will include spirometry, lung volumes, and DLCO.

Genetic Counseling Visit (Optional):

Should you be interested in having a visit with a genetic counselor associated with the research team, a standard new patient visit with the counselor can be arranged with your first visit for the study, or at a follow-up visit. The study will pay for one visit with the genetic counselor, who will provide a standard session that is tailored to your and your family's history. Some of the information obtained during the visit may be used in this research study, to help us understand the counselling needs of relatives of patients with pulmonary fibrosis. The counselor may discuss aspects of clinical care, including clinical genetic testing. The study will not pay for clinical genetic testing, but the genetic counselor will discuss when clinical genetic testing is appropriate and which family members are most informative to undergo clinical genetic testing.

Specimen collection, processing, and banking: Each subject will have 50 ml blood collected on enrollment and on the day of repeat HRCT. Lymphocytes will be saved for generation of lymphoblastoid cells, DNA isolation, and telomere length analysis. Both serum and plasma will be saved for further studies.

ELIGIBILITY:
Eligibility Requirements:

1. Bloodline members of an affected individual from a family in which two or more members of a family are known to have Idiopathic Interstitial Pneumonia (IIP) and who have no personal diagnosis of IIP or IPF
2. Sibling or adult child of an affected individual

Exclusion Criteria:

1. Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by the IRB).
2. Inability to travel to Nashville for 1-2 outpatient visits and/or complete a written or online version of the Interstitial Lung Disease Questionnaire
3. Age < 40 or >75 years old. If the affected relative was younger than 50 years old at the time of IIP diagnosis, potential subjects between age 18 and 40 years may participate when they are up to 10 years younger than the age at relative's diagnosis.
4. Underlying disease with signs and symptoms that could be confused with IIP or IPF symptoms (i.e., rheumatoid arthritis or other connective tissue diseases, occupational lung disease, chemotherapy, etc.)
5. Thought to be unsuitable for participation in the study in the opinion of the investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1) Bloodline members of an affected individual from a family in which two or more members of a family bloodline are known to have had proven Idiopathic Interstitial Pneumonia (IIP) and who have no known diagnosis of IIP or IPF
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
clinical diagnosis of interstitial lung disease | Until anticipated study completion of 01-30-2030
  by ATS/ERS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Salisbury, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States